CLINICAL TRIAL: NCT01187212
Title: A Randomized Phase II Study of Capecitabine and Cisplatin (XP) +/- Sorafenib (Nexavar®) in Patients With Advanced Gastric Cancer
Brief Title: Sorafenib Trial in Advanced and/or Recurrent Gastric Adenocarcinoma: Treatment Evaluation: STARGATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMC1002
Record Dates: First submitted 2010-08-19; First posted 2010-08-24 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Malignant Neoplasm of Stomach; Effects of Chemotherapy
Keywords: First line chemotherapy in advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capecitabine/Cisplatin (Active Comparator): Capecitabine 1000 milligram (mg) / m² po bid (D1-14) Cisplatin 80 mg / m² IV Day (D) 1
  Interventions: Drug: Capecitabine/Cisplatin
- Capecitabine/Cisplatin + Sorafenib (Experimental): Capecitabine 800 mg / m² po bid (D1-14) Cisplatin 60 mg / m² IV Day 1 Sorafenib 400 mg p.o. bid continuous dosing
  Interventions: Drug: Capecitabine/Cisplatin + Sorafenib

INTERVENTIONS:
Drug: Capecitabine/Cisplatin + Sorafenib — Capecitabine 800 mg / m² po bid (D1-14) Cisplatin 60 mg / m² IV Day 1 Sorafenib 400 mg p.o. bid continuous dosing
  Other Names: Xeloda; Nexavar
  Arms: Capecitabine/Cisplatin + Sorafenib
Drug: Capecitabine/Cisplatin — Capecitabine 1000 milligram (mg) / m² po bid (D1-14) Cisplatin 80 mg / m² IV Day 1
  Other Names: Xeloda
  Arms: Capecitabine/Cisplatin

SUMMARY:
This study investigates the efficacy and safety profiles of sorafenib in combination of capecitabine and cisplatin, one of standard chemotherapy regimens in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Histological or cytological documentation of gastric adenocarcinoma or gastroesophageal junction adenocarcinoma.;
3. Metastatic gastric adenocarcinoma or metastatic gastroesophageal junction adenocarcinoma, initially diagnosed or recurrent.
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors
5. ECOG Performance Status of 0 or 1
6. Life expectancy of at least 3 months
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

   * Hemoglobin ≥ 9.0 g / dl
   * Absolute neutrophil count (ANC) ≥1,500 / mm3
   * Platelet count ≥ 100,000 / mm3
   * Total bilirubin < 1.5 x upper limit of normal
   * ALT and AST < 2.5 x upper limit of normal (< 5 x ULN for patients with liver involvement of their cancer)
   * International normalized ratio of PT (PT-INR) / PTT < 1.5 x ULN
8. Creatinine Clearance ≥ 60 ml / min (based on Cockcroft and Gault formula)
9. Ability to understand and willingness to sign a written informed consent. Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

1. Patients with local-regional gastric or gastroesophageal adenocarcinoma (no para-aortic nodes or visceral structure-invading primary [T4]) who can potentially become candidates for surgery with curative intent following systemic therapy
2. History of cardiac disease:

   * Congestive heart failure >NYHA class 2; unstable angina (angina symptoms present at rest), new-onset angina (began within last three months prior to randomization) or myocardial infarction within six months prior to randomization;
   * Ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted);
   * Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg) despite optimal medical management
3. Past or concurrent history of neoplasm < 5 years prior to start of study treatment other than gastric adenocarcinoma or gastroesophageal junction adenocarcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix uteri or superficial bladder tumors [Ta noninvasive tumor (Ta), carcinoma in situ (Tis) and T1 (tumor invades lamina propria)]
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization
5. Evidence of gastrointestinal perforation or bowel obstruction during the screening period
6. Evidence or history of bleeding diathesis or coagulopathy
7. Non-healing wound, ulcer, or bone fracture
8. History of gastrointestinal bleeding > grade 1 CTCAE version 4.0 within 4 weeks prior to randomization
9. History of any other bleeding > grade 2 according to CTCAE version 4.0 within 4 weeks prior to randomization
10. Known psychiatric and neurological disorders including known peripheral or autonomous neuropathy or hearing impairment > grade 1 according to CTCAE version 4.0

    * However, if the patient already has known irreversible grade 4 hearing loss (>90 decibels (dB) bilaterally) at baseline, he or she is eligible at the investigator's discretion
11. Pregnant or lactating women, women of childbearing potential not employing adequate contraception [Women of childbearing potential must have a negative serum pregnancy test performed within seven days prior to the start of treatment. Of note, both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and four weeks after the completion of trial or 6 months after last dose of cisplatin (whichever is greater). The definition of effective contraception will be based on the clinical judgment of the principal investigator or a designated associate.]
12. Evidence of infection (> grade 2 )
13. History of HIV infection or chronic / active hepatitis B or C
14. Evidence of brain metastasis. Patients with unexplained neurological symptoms will undergo a CT scan or MRI of the brain to exclude metastases.
15. Seizure disorder requiring treatment with medications that affect CYP 3A4
16. History of organ allograft
17. Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes or excipients in the formulation given during the course of this trial
18. Any condition that is unstable or could jeopardize the safety of the patient and his / her compliance in the study
19. Inability to swallow or retain oral medications
20. Any malabsorption condition that the investigator deems would jeopardize the absorption or pharmacokinetics of the study medication
21. Uncorrected dehydration
22. Known dihydropyrimidine dehydrogenase deficiency
23. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
24. Evidence of thrombotic or embolic disease, including cerebrovascular accident, transient ischemic attacks, or pulmonary embolus within the past 6 months
25. Any tumor with characteristics that the investigator deems unsuitable for potentially cytoreductive therapy due to likelihood of severe bleeding or perforation such as ulcerations or hemorrhage. Excluded therapies and medications
26. Prior or concomitant systemic anticancer therapy including cytotoxic therapy, targeted agents, or experimental therapy for gastric cancer. However, (neo)-adjuvant cytotoxic therapy is permitted if the last dose was administered > 6 months (12 months for platinum based therapy) before start of study medication in this study.
27. Radiotherapy prior to or during the study (palliative radiotherapy will be allowed as described in the 'prior and concomitant therapy section',4.3.7)
28. Use of biologic response modifiers, such as granulocyte G-CSF, within 3 weeks of study entry and during the study.
29. Investigational drug therapy outside of this trial during or within 4 weeks prior to randomization
30. Previous exposure to a Ras pathway inhibitor such MEK or Raf inhibitors or any farnesyl transferase inhibitors
31. Therapeutic anticoagulation with vitamin K antagonists such as warfarin, or with heparins or heparinoids

    * Low dose warfarin (1 mg p.o. q.d.) is permitted if the international normalized ratio is < 1.5
    * Low-dose aspirin is permitted (≤ 100 mg daily)
    * Prophylactic doses of heparin are permitted
    * For patients on warfarin, the INR will be measured prior to initiation of sorafenib, and patients will be monitored regularly for changes in prothrombin time, INR or clinical bleeding episodes as infrequent bleeding or elevations in the INR have been reported in some patients taking warfarin while on sorafenib therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Best tumor response | 2 years
Duration of response | 2 years
Disease control rate | 2 years
Safety profiles | up to 2years
  Toxicity profiles will be assessed with the patient 30 +/- 3 days after the last intake of study medication is required.
Best tumoral response of 2nd line sorafenib | 2 years
  Best tumoral response of sorafenib in patients who progressed on capecitabine and cisplatin (control group)
Progression-free survival of 2nd line sorafenib | 2years
  Progression-free survival of sorafenib in patients who progressed on capecitabine and cisplatin (control group)
Biomarker for sorafenib | 2years
  Blood and tumor tissue will be collected during the study, and analyzed for biomarker at the end of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yoon-Koo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Ahn YO, Park BJ, Yoo KY, Kim NK, Heo DS, Lee JK, Ahn HS, Kang DH, Kim H, Lee MS, et al. Incidence estimation of stomach cancer among Koreans. J Korean Med Sci. 1991 Mar;6(1):7-14. doi: 10.3346/jkms.1991.6.1.7. PMID 1888453
- [Background] Bang YJ, Kang WK, Kang YK, Kim HC, Jacques C, Zuber E, Daglish B, Boudraa Y, Kim WS, Heo DS, Kim NK. Docetaxel 75 mg/m(2) is active and well tolerated in patients with metastatic or recurrent gastric cancer: a phase II trial. Jpn J Clin Oncol. 2002 Jul;32(7):248-54. doi: 10.1093/jjco/hyf057. PMID 12324575
- [Background] Borgstrom P, Gold DP, Hillan KJ, Ferrara N. Importance of VEGF for breast cancer angiogenesis in vivo: implications from intravital microscopy of combination treatments with an anti-VEGF neutralizing monoclonal antibody and doxorubicin. Anticancer Res. 1999 Sep-Oct;19(5B):4203-14. PMID 10628376
- [Background] Bremnes RM, Camps C, Sirera R. Angiogenesis in non-small cell lung cancer: the prognostic impact of neoangiogenesis and the cytokines VEGF and bFGF in tumours and blood. Lung Cancer. 2006 Feb;51(2):143-58. doi: 10.1016/j.lungcan.2005.09.005. Epub 2005 Dec 19. PMID 16360975
- [Background] Chong G, Cunningham D. Gastrointestinal cancer: recent developments in medical oncology. Eur J Surg Oncol. 2005 Jun;31(5):453-60. doi: 10.1016/j.ejso.2005.02.026. Epub 2005 Apr 13. PMID 15922879
- [Background] Constenla M, Garcia-Arroyo R, Lorenzo I, Carrete N, Campos B, Palacios P. Docetaxel, 5-fluorouracil, and leucovorin as treatment for advanced gastric cancer: results of a phase II study. Gastric Cancer. 2002;5(3):142-7. doi: 10.1007/s101200200025. PMID 12378340
- [Background] Einzig AI, Neuberg D, Remick SC, Karp DD, O'Dwyer PJ, Stewart JA, Benson AB 3rd. Phase II trial of docetaxel (Taxotere) in patients with adenocarcinoma of the upper gastrointestinal tract previously untreated with cytotoxic chemotherapy: the Eastern Cooperative Oncology Group (ECOG) results of protocol E1293. Med Oncol. 1996 Jun;13(2):87-93. doi: 10.1007/BF02993858. PMID 9013471
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Graziano F, Catalano V, Baldelli AM, Giordani P, Testa E, Lai V, Catalano G, Battelli N, Cascinu S. A phase II study of weekly docetaxel as salvage chemotherapy for advanced gastric cancer. Ann Oncol. 2000 Oct;11(10):1263-6. doi: 10.1023/a:1008373814453. PMID 11106114
- [Background] Jain RK. Normalizing tumor vasculature with anti-angiogenic therapy: a new paradigm for combination therapy. Nat Med. 2001 Sep;7(9):987-9. doi: 10.1038/nm0901-987. No abstract available. PMID 11533692
- [Background] Kamiyama M, Ichikawa Y, Ishikawa T, Chishima T, Hasegawa S, Hamaguchi Y, Nagashima Y, Miyagi Y, Mitsuhashi M, Hyndman D, Hoffman RM, Ohki S, Shimada H. VEGF receptor antisense therapy inhibits angiogenesis and peritoneal dissemination of human gastric cancer in nude mice. Cancer Gene Ther. 2002 Feb;9(2):197-201. doi: 10.1038/sj.cgt.7700428. PMID 11857038
- [Background] Kanai T, Konno H, Tanaka T, Baba M, Matsumoto K, Nakamura S, Yukita A, Asano M, Suzuki H, Baba S. Anti-tumor and anti-metastatic effects of human-vascular-endothelial-growth-factor-neutralizing antibody on human colon and gastric carcinoma xenotransplanted orthotopically into nude mice. Int J Cancer. 1998 Sep 11;77(6):933-6. doi: 10.1002/(sici)1097-0215(19980911)77:63.0.co;2-0. PMID 9714067
- [Background] Kang YK, Kang WK, Shin DB, Chen J, Xiong J, Wang J, Lichinitser M, Guan Z, Khasanov R, Zheng L, Philco-Salas M, Suarez T, Santamaria J, Forster G, McCloud PI. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin as first-line therapy in patients with advanced gastric cancer: a randomised phase III noninferiority trial. Ann Oncol. 2009 Apr;20(4):666-73. doi: 10.1093/annonc/mdn717. Epub 2009 Jan 19. PMID 19153121
- [Background] Karayiannakis AJ, Syrigos KN, Polychronidis A, Zbar A, Kouraklis G, Simopoulos C, Karatzas G. Circulating VEGF levels in the serum of gastric cancer patients: correlation with pathological variables, patient survival, and tumor surgery. Ann Surg. 2002 Jul;236(1):37-42. doi: 10.1097/00000658-200207000-00007. PMID 12131083
- [Background] Kawasaki T, Kitsukawa T, Bekku Y, Matsuda Y, Sanbo M, Yagi T, Fujisawa H. A requirement for neuropilin-1 in embryonic vessel formation. Development. 1999 Nov;126(21):4895-902. doi: 10.1242/dev.126.21.4895. PMID 10518505
- [Background] Kitsukawa T, Shimono A, Kawakami A, Kondoh H, Fujisawa H. Overexpression of a membrane protein, neuropilin, in chimeric mice causes anomalies in the cardiovascular system, nervous system and limbs. Development. 1995 Dec;121(12):4309-18. doi: 10.1242/dev.121.12.4309. PMID 8575331
- [Background] Lackner C, Jukic Z, Tsybrovskyy O, Jatzko G, Wette V, Hoefler G, Klimpfinger M, Denk H, Zatloukal K. Prognostic relevance of tumour-associated macrophages and von Willebrand factor-positive microvessels in colorectal cancer. Virchows Arch. 2004 Aug;445(2):160-7. doi: 10.1007/s00428-004-1051-z. Epub 2004 Jun 30. PMID 15232739
- [Background] Maeda K, Chung YS, Ogawa Y, Takatsuka S, Kang SM, Ogawa M, Sawada T, Sowa M. Prognostic value of vascular endothelial growth factor expression in gastric carcinoma. Cancer. 1996 Mar 1;77(5):858-63. doi: 10.1002/(sici)1097-0142(19960301)77:53.0.co;2-a. PMID 8608475
- [Background] Mai M, Sakata Y, Kanamaru R, Kurihara M, Suminaga M, Ota J, Hirabayashi N, Taguchi T, Furue H. [A late phase II clinical study of RP56976 (docetaxel) in patients with advanced or recurrent gastric cancer: a cooperative study group trial (group B)]. Gan To Kagaku Ryoho. 1999 Mar;26(4):487-96. Japanese. PMID 10097745
- [Background] Mavroudis D, Kourousis C, Androulakis N, Kalbakis K, Agelaki S, Kakolyris S, Souglakos J, Sarra E, Vardakis N, Hatzidaki D, Sarmonis G, Georgoulias V. Frontline treatment of advanced gastric cancer with docetaxel and granulocyte colony-stimulating factor (G-CSF): a phase II trial. Am J Clin Oncol. 2000 Aug;23(4):341-4. doi: 10.1097/00000421-200008000-00005. PMID 10955859
- [Background] McCarty MF, Wey J, Stoeltzing O, Liu W, Fan F, Bucana C, Mansfield PF, Ryan AJ, Ellis LM. ZD6474, a vascular endothelial growth factor receptor tyrosine kinase inhibitor with additional activity against epidermal growth factor receptor tyrosine kinase, inhibits orthotopic growth and angiogenesis of gastric cancer. Mol Cancer Ther. 2004 Sep;3(9):1041-8. PMID 15367698
- [Background] Moreira IS, Fernandes PA, Ramos MJ. Vascular endothelial growth factor (VEGF) inhibition--a critical review. Anticancer Agents Med Chem. 2007 Mar;7(2):223-45. doi: 10.2174/187152007780058687. PMID 17348829
- [Background] Oh SY, Kwon HC, Kim SH, Jang JS, Kim MC, Kim KH, Han JY, Kim CO, Kim SJ, Jeong JS, Kim HJ. Clinicopathologic significance of HIF-1alpha, p53, and VEGF expression and preoperative serum VEGF level in gastric cancer. BMC Cancer. 2008 May 1;8:123. doi: 10.1186/1471-2407-8-123. PMID 18452596
- [Background] Otrock ZK, Makarem JA, Shamseddine AI. Vascular endothelial growth factor family of ligands and receptors: review. Blood Cells Mol Dis. 2007 May-Jun;38(3):258-68. doi: 10.1016/j.bcmd.2006.12.003. Epub 2007 Mar 6. PMID 17344076
- [Background] Raspollini MR, Amunni G, Villanucci A, Baroni G, Boddi V, Taddei GL. Prognostic significance of microvessel density and vascular endothelial growth factor expression in advanced ovarian serous carcinoma. Int J Gynecol Cancer. 2004 Sep-Oct;14(5):815-23. doi: 10.1111/j.1048-891X.2004.014514.x. PMID 15361189
- [Background] Ridwelski K, Gebauer T, Fahlke J, Kroning H, Kettner E, Meyer F, Eichelmann K, Lippert H. Combination chemotherapy with docetaxel and cisplatin for locally advanced and metastatic gastric cancer. Ann Oncol. 2001 Jan;12(1):47-51. doi: 10.1023/a:1008328501128. PMID 11249048
- [Background] Roth AD, Maibach R, Martinelli G, Fazio N, Aapro MS, Pagani O, Morant R, Borner MM, Herrmann R, Honegger H, Cavalli F, Alberto P, Castiglione M, Goldhirsch A. Docetaxel (Taxotere)-cisplatin (TC): an effective drug combination in gastric carcinoma. Swiss Group for Clinical Cancer Research (SAKK), and the European Institute of Oncology (EIO). Ann Oncol. 2000 Mar;11(3):301-6. doi: 10.1023/a:1008342013224. PMID 10811496
- [Background] Shah MA, Ramanathan RK, Ilson DH, Levnor A, D'Adamo D, O'Reilly E, Tse A, Trocola R, Schwartz L, Capanu M, Schwartz GK, Kelsen DP. Multicenter phase II study of irinotecan, cisplatin, and bevacizumab in patients with metastatic gastric or gastroesophageal junction adenocarcinoma. J Clin Oncol. 2006 Nov 20;24(33):5201-6. doi: 10.1200/JCO.2006.08.0887. PMID 17114652
- [Background] Simiantonaki N, Taxeidis M, Jayasinghe C, Kirkpatrick CJ. Epithelial expression of VEGF receptors in colorectal carcinomas and their relationship to metastatic status. Anticancer Res. 2007 Sep-Oct;27(5A):3245-50. PMID 17970067
- [Background] Song ZJ, Gong P, Wu YE. Relationship between the expression of iNOS,VEGF,tumor angiogenesis and gastric cancer. World J Gastroenterol. 2002 Aug;8(4):591-5. doi: 10.3748/wjg.v8.i4.591. PMID 12174362
- [Background] Sulkes A, Smyth J, Sessa C, Dirix LY, Vermorken JB, Kaye S, Wanders J, Franklin H, LeBail N, Verweij J. Docetaxel (Taxotere) in advanced gastric cancer: results of a phase II clinical trial. EORTC Early Clinical Trials Group. Br J Cancer. 1994 Aug;70(2):380-3. doi: 10.1038/bjc.1994.310. PMID 7914428
- [Background] Sutter AP, Zeitz M, Scherubl H. Recent results in understanding molecular pathways in the medical treatment of esophageal and gastric cancer. Onkologie. 2004 Feb;27(1):17-21. doi: 10.1159/000075600. PMID 15007244
- [Background] Sweeney CJ, Miller KD, Sissons SE, Nozaki S, Heilman DK, Shen J, Sledge GW Jr. The antiangiogenic property of docetaxel is synergistic with a recombinant humanized monoclonal antibody against vascular endothelial growth factor or 2-methoxyestradiol but antagonized by endothelial growth factors. Cancer Res. 2001 Apr 15;61(8):3369-72. PMID 11309294
- [Background] Sym SJ, Chang HM, Ryu MH, Lee JL, Kim TW, Yook JH, Oh ST, Kim BS, Kang YK. Neoadjuvant docetaxel, capecitabine and cisplatin (DXP) in patients with unresectable locally advanced or metastatic gastric cancer. Ann Surg Oncol. 2010 Apr;17(4):1024-32. doi: 10.1245/s10434-009-0838-1. Epub 2009 Nov 26. PMID 19941081
- [Background] Takahashi Y, Cleary KR, Mai M, Kitadai Y, Bucana CD, Ellis LM. Significance of vessel count and vascular endothelial growth factor and its receptor (KDR) in intestinal-type gastric cancer. Clin Cancer Res. 1996 Oct;2(10):1679-84. PMID 9816116
- [Background] Tanigawa N, Amaya H, Matsumura M, Shimomatsuya T, Horiuchi T, Muraoka R, Iki M. Extent of tumor vascularization correlates with prognosis and hematogenous metastasis in gastric carcinomas. Cancer Res. 1996 Jun 1;56(11):2671-6. PMID 8653715
- [Background] Tas F, Duranyildiz D, Oguz H, Camlica H, Yasasever V, Topuz E. Circulating serum levels of angiogenic factors and vascular endothelial growth factor receptors 1 and 2 in melanoma patients. Melanoma Res. 2006 Oct;16(5):405-11. doi: 10.1097/01.cmr.0000222598.27438.82. PMID 17013089
- [Background] Tsutsui S, Kume M, Era S. Prognostic value of microvessel density in invasive ductal carcinoma of the breast. Breast Cancer. 2003;10(4):312-9. doi: 10.1007/BF02967651. PMID 14634509
- [Background] Van Cutsem E, Moiseyenko VM, Tjulandin S, Majlis A, Constenla M, Boni C, Rodrigues A, Fodor M, Chao Y, Voznyi E, Risse ML, Ajani JA; V325 Study Group. Phase III study of docetaxel and cisplatin plus fluorouracil compared with cisplatin and fluorouracil as first-line therapy for advanced gastric cancer: a report of the V325 Study Group. J Clin Oncol. 2006 Nov 1;24(31):4991-7. doi: 10.1200/JCO.2006.06.8429. PMID 17075117
- [Background] Wang G, Dong Z, Xu G, Yang Z, Shou C, Wang N, Liu T. The effect of antibody against vascular endothelial growth factor on tumor growth and metastasis. J Cancer Res Clin Oncol. 1998;124(11):615-20. doi: 10.1007/s004320050223. PMID 9860290
- [Background] Wang TB, Deng MH, Qiu WS, Dong WG. Association of serum vascular endothelial growth factor-C and lymphatic vessel density with lymph node metastasis and prognosis of patients with gastric cancer. World J Gastroenterol. 2007 Mar 28;13(12):1794-7; discussion 1797-8. doi: 10.3748/wjg.v13.i12.1794. PMID 17465468
- [Background] Whitaker GB, Limberg BJ, Rosenbaum JS. Vascular endothelial growth factor receptor-2 and neuropilin-1 form a receptor complex that is responsible for the differential signaling potency of VEGF(165) and VEGF(121). J Biol Chem. 2001 Jul 6;276(27):25520-31. doi: 10.1074/jbc.M102315200. Epub 2001 May 1. PMID 11333271
- [Background] Yamamoto S, Yasui W, Kitadai Y, Yokozaki H, Haruma K, Kajiyama G, Tahara E. Expression of vascular endothelial growth factor in human gastric carcinomas. Pathol Int. 1998 Jul;48(7):499-506. doi: 10.1111/j.1440-1827.1998.tb03940.x. PMID 9701011